CLINICAL TRIAL: NCT02334319
Title: A Molecularly Driven Pilot Study of Preoperative Ganetespib in Resectable Squamous Cell Carcinoma of the Head and Neck (SCCHN)
Brief Title: Ganetespib Window of Opportunity Study in Head and Neck Cancers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Emory University (Other)
Collaborators: Synta Pharmaceuticals Corp. (Industry)
Responsible Party: Principal Investigator, Nabil F. Saba, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00070264; WINSHIP2572-13 (Registry Identifier: Emory University/Winship Cancer Institute); NCI-2014-02605 (Other: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2015-01-06; First posted 2015-01-08 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Stage I Hypopharyngeal Squamous Cell Carcinoma; Stage I Laryngeal Squamous Cell Carcinoma; Stage I Oral Cavity Squamous Cell Carcinoma; Stage I Oropharyngeal Squamous Cell Carcinoma; Stage II Hypopharyngeal Squamous Cell Carcinoma; Stage II Laryngeal Squamous Cell Carcinoma; Stage II Oral Cavity Squamous Cell Carcinoma; Stage II Oropharyngeal Squamous Cell Carcinoma; Stage III Hypopharyngeal Squamous Cell Carcinoma; Stage III Laryngeal Squamous Cell Carcinoma; Stage III Oral Cavity Squamous Cell Carcinoma; Stage III Oropharyngeal Squamous Cell Carcinoma; Stage IVA Hypopharyngeal Squamous Cell Carcinoma; Stage IVA Laryngeal Squamous Cell Carcinoma; Stage IVA Oral Cavity Squamous Cell Carcinoma; Stage IVA Oropharyngeal Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — STA 9090

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (ganetespib, surgery) (Experimental): Patients receive ganetespib IV over 1 hour twice weekly for 2 weeks in the absence of disease progression or unacceptable toxicity. Patients then undergo surgery the day after the last dose of ganetespib.
  Interventions: Drug: Ganetespib; Procedure: Therapeutic Conventional Surgery; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Ganetespib — Given IV
  Other Names: Hsp90 Inhibitor STA-9090; STA-9090
Procedure: Therapeutic Conventional Surgery — Undergo surgery
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This pilot clinical trial studies how well ganetespib works before surgery in treating patients with stage I-IVA squamous cell carcinoma of the head and neck that can be removed by surgery. Ganetespib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Studying samples of blood and tissue in the laboratory from patients receiving ganetespib may help doctors learn more about the effects of ganetespib on cells. It may also help doctors understand how well patients respond to treatment.

DETAILED DESCRIPTION:
Ganetespib is a small molecule inhibitor of HSP90 that is currently being studied in several ongoing clinical trials. Investigators have demonstrated that ganetespib sensitizes colorectal cell lines to the effects of chemo radiotherapy in vitro. Ganetespib may have an anti-tumor effect in head and neck cancer. The investigators propose this pilot study as a first step to examine the activity of ganetespib in patients with locally advanced squamous cell carcinoma of the head and neck (SCCHN) who have a planned surgical resection.

Ganetespib has not been investigated in SCCHN. This protocol is a window of opportunity trial that will be looking at whether there is a rationale for pursuing this agent in future development of clinical trials that would then focus on therapeutic interventions with or without radiotherapy. There are therefore no clinical trials currently opened using ganetespib in SCCHN and listed on ClinicalTrials.gov. It is not clear if patients who receive this drug prior to surgery will benefit from this intervention.

In this study, ganetespib will be administered twice weekly (doses approximately 72 hours apart) for 2 weeks, followed by surgery the day after the last dose of the study drug. There will be 3 dose levels, 80, 100 and 150mg/m² as highest dose. These doses were chosen based on the following considerations. In a Phase 1 study (protocol 9090-01) investigating a twice-weekly ganetespib treatment schedule, doses up to 173 mg/m² were well tolerated, with manageable diarrhea and fatigue being the most common adverse events. Extensive correlative studies and pharmacokinetic (PK)/pharmacodynamic (PD) modeling of preclinical data suggest that in humans the effective dose range for ganetespib is 70-150 mg/m². Therefore, 80 mg/m² is within the range of ganetespib effectiveness and 150 mg/m² twice weekly is a well-tolerated dose.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have pathologically-confirmed, resectable, squamous cell carcinoma of the oral cavity, oropharynx, larynx or hypopharynx
* Disease may be stage I, II, III or IVa (as long as it is deemed resectable by the surgical team)
* Tumor must be surgically resectable and curable with conventional surgery
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Patients must give documented informed consent to participate in this study
* Absolute-neutrophil count (ANC) ≥ 1500/mm³
* Platelet count ≥ 100,000/mm³
* Total bilirubin ≤ within upper limit of normal (ULN)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 x ULN
* Creatinine ≤ 1.5 x ULN
* Lipase levels < 1.5 x ULN
* Amylase levels < 1.5 x ULN

Exclusion Criteria:

* Prior therapy with a known heat shock protein 90 (HSP90) inhibitor
* Poor venous access for study drug administration; in this case, patients would require a peripheral or central indwelling catheter for study drug administration; study drug administration via indwelling catheters is prohibited at this time unless silicone based catheters are used; anything other than catheters made from silicone are not allowed with ganetespib therapy
* History of severe allergic or hypersensitivity reactions to excipients (e.g., polyethylene glycol [PEG] 300 and polysorbate 80)
* Treatment with chronic immunosuppressant (e.g., cyclosporine following transplantation)
* Uncontrolled undercurrent illness including, but not limited to, human immunodeficiency virus (HIV)-positive subjects receiving combination antiretroviral therapy, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, ventricular arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Other medications, or severe acute/chronic medical or psychiatric condition, or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the subject inappropriate for entry into this study
* Documented evidence of distant metastases or brain metastases
* Active malignancy besides head and neck squamous cell cancer (HNSCC) or primary skin basal cell carcinoma; (patients with a concomitant malignancy that has not progressed within 12 months of study entry are eligible)
* History of documented congestive heart failure (CHF), New York Heart Association class II/III/IV, with a history of dyspnea, orthopnea or edema that requires current treatment with angiotensin converting enzyme inhibitors, angiotensin II receptor blockers, beta-blockers or diuretics; NOTE: use of these medications for the treatment of hypertension is allowed
* Peripheral neuropathy that is grade 2 or higher
* Pregnancy or lactation; patients of child bearing age must agree to use adequate contraception
* Patients residing in prison
* CARDIAC EXCLUSION CRITERIA:

  * Known serious cardiac illness or medical conditions, including but not limited to:

    * Clinically unstable cardiac disease, including unstable atrial fibrillation, symptomatic bradycardia, unstable congestive heart failure, active myocardial ischemia, or indwelling temporary pacemaker
    * Ventricular tachycardia or a supraventricular tachycardia that requires treatment with a class Ia antiarrhythmic drug (e.g., quinidine, procainamide, disopyramide) or class III antiarrhythmic drug (e.g., sotalol, amiodarone, dofetilide); use of other antiarrhythmic drugs is permitted
    * Use of medications that have been linked to the occurrence of Torsades de pointes
    * Second- or third-degree atrioventricular (AV) block unless treated with a permanent pacemaker
    * Complete left bundle branch block (LBBB)
    * History of long QT syndrome or a family member with this condition
    * Corrected QT (QTc) > 470 ms (average of triplicate electrocardiogram [ECG] recordings); a consistent method of QTc calculation must be used for each patient's QTc measurements; QTcF (Fridericia's formula) is preferred
    * Serum potassium, magnesium, or calcium levels in the following ranges:

      * Potassium < 3.4 or > 5.1 mmol/L
      * Magnesium < 1.4 or > 2.4 mg/dL
      * Calcium < 8.9 or > 10.5 mg/dL

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-12; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Change in expression of biomarkers in tissue samples, assessed by immunohistochemistry (IHC) | Baseline to up to 24 months
  The biomarker expression of pre-, post-treatment, and their change will be described by summary statistics along with 95% confidence interval (CI) for the estimated mean. A paired sample Wilcoxon signed rank test will be considered to test whether the mean of post-treatment expression is different from the pre-treatment expression. This analysis will be done separately by each of the three dose levels, and by pooling all dose levels together. Kruskal-Wallis test will also be carried out.
Change in biomarker expression in blood samples | Baseline to up to 24 months
  The biomarker expression of pre-, post-treatment, as well as their change will be described by summary statistics along with 95% CI for the estimated mean. A paired sample Wilcoxon signed rank test will be considered to test whether the mean of post-treatment expression is different from that of the pre-treatment expression. This analysis will be done separately by each of the three dose levels, as well as by pooling all dose levels together. Kruskal-Wallis test will also be carried out.

CONTACTS AND LOCATIONS:
Overall Officials: Nabil F. Saba, MD, Principal Investigator — Emory University/Winship Cancer Institute
Locations (2):
- United States (2):
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University/Winship Cancer Institute, Atlanta, Georgia